CLINICAL TRIAL: NCT05594225
Title: Tele-Rehabilitation to Improve Mild Traumatic Brain Injury Recovery and Reduce Subsequent Injury Risk
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Binghamton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-1352
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Participants will enroll and undergo initial testing within three weeks of mTBI, be randomized to an 8-week vNDTT or standard-of-care intervention, return for post-intervention testing, and be monitored for subsequent MSK injuries in the three months after mTBI
Who Masked: Outcomes Assessor
Masking Description: The study PI, Co-Is, and the biostatistician will not know group assignments until after the primary analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Neuromuscular/Dual-Task Training (Experimental): The vNDTT strategy incorporates lower body strength exercises with landing stabilization focus. Exercises will begin after the initial study visit and last for 8 weeks.
  Interventions: Behavioral: Virtual Neuromuscular/Dual-Task Training
- Standard-of-care (No Intervention): Participants will be provided routine instructions related to physical activity and rehabilitation exercises

INTERVENTIONS:
Behavioral: Virtual Neuromuscular/Dual-Task Training — The vNDTT strategy incorporates lower body strength exercises with landing stabilization focus. Exercises will begin after the initial study visit and last for 8 weeks.
  Arms: Virtual Neuromuscular/Dual-Task Training

SUMMARY:
The goal of this clinical trial is to examine the feasibility, utility, and efficacy of a smartphone-based assessment battery and remotely administered virtual Neuromuscular/Dual-Task (vNDT) intervention among healthy U.S. military service members and physically active young adults with a recent concussion.

DETAILED DESCRIPTION:
Aim 1. Determine the baseline neuromuscular/dual-task performance characteristics among a sample of active-duty military service members compared to physically active young adult civilians.

The investigators hypothesize that active-duty military service members will have similar baseline gait and dual-task abilities as civilians, demonstrating translation potential between populations.

The investigators also hypothesize that baseline gait and dual-task abilities will be influenced by history of prior mTBI injuries among military Service Members.

Aim 2. Examine the efficacy of a smartphone-based vNDTT intervention to reduce musculoskeletal injury and improve neuromuscular/dual-task performance after a recent mTBI.

The investigators hypothesize that those randomized to the intervention within three weeks of mTBI will have a lower risk of MSK injury in the 3-month period following mTBI, relative to standard-of-care.

The investigators also hypothesize that those randomized to the intervention within three weeks of mTBI will have better post-intervention gait and dual-task performance than those assigned to standard-of-care, despite similar baseline performance.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age at the time of enrollment
* Mild TBI or concussion diagnosis by a physician
* Confirmed MTBI diagnosis via VA/DOD guidelines at time of enrollment
* Participation in regular physical activity prior to injury (confirmed via the Global Physical Activity Questionnaire [GPAQ]) (Cleland et al., 2014; Keating et al., 2019)
* Access to a smartphone for app download

Exclusion Criteria:

* Moderate or severe TBI
* Pre-injury neurological disorder
* Abnormal brain imaging findings (if performed as a part of routine care)
* Previous TBI (mild/moderate/severe) <12 months prior to enrollment other than the current injury for which they are being seen

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Injury rate | 3 months after mTBI
  Acute musculoskeletal injury rate

SECONDARY OUTCOMES:
Intervention adherence | Upon enrollment and for the subsequent 8 weeks
  Virtually logging a training session on the smartphone application (# of sessions logged/planned sessions
Quality of Life Domains: Mobility, Depressive Symptoms, Fatigue, Pain Interference | During the initial (post-injury) evaluation and again at the follow-up (8 weeks after initial evaluation) test
  Patient-Reported Outcomes Measurement Information System (PROMIS) global questionnaire
Sleep quality | During the initial (post-injury) evaluation and again at the follow-up (8 weeks after initial evaluation) test
  Participants will complete the Pittsburgh Sleep Quality Inventory
Dizziness | During the initial (post-injury) evaluation and again at the follow-up (8 weeks after initial evaluation) test
  Participants will complete the Dizziness Handicap Inventory
Anxiety | During the initial (post-injury) evaluation and again at the follow-up (8 weeks after initial evaluation) test
  Participants will complete the General Anxiety Disorder - 7 scale
Single/dual-task standing and gait | During the initial (post-injury) evaluation and again at the follow-up (8 weeks after initial evaluation) test
  Participants will perform walking trials under single and dual-task conditions

CONTACTS AND LOCATIONS:
Overall Officials: David R Howell, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified/blinded IPD data may be made available upon reasonable request.